CLINICAL TRIAL: NCT00206557
Title: The Use of Selective Estrogen Receptor Modulators in the Treatment of Schizophrenia- a Pilot Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Alfred (Other)
Collaborators: Stanley Medical Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APRC 146/02; 03T-422
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2007-04-23 (Estimated); Status verified 2007-04

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorder
Keywords: Schizophrenia; Mental Illness; Hormone Therapy; Post-menopausal; SERM; Raloxifene
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Mental Disorders | interventions — Raloxifene Hydrochloride; Estradiol

INTERVENTIONS:
Drug: Raloxifene
Drug: Estradiol/dyhydroprogestrone

SUMMARY:
The aim of the project is to investigate the use of raloxifene (a new form of estrogen) as a treatment for schizophrenia in postmenopausal women. Raloxifene is a selective estrogen receptor modulator (SERM) which means that it can affect the central nervous system effects of estrogen (eg: improving emotional symptoms, memory, information processing and concentration), without adversely affecting reproductive tissue / organs such as breast, uterus and ovaries.We are conducting a double blind placebo controlled 3 month duration study comparing the psychotic symptom response between three groups of postmenopausal women with schizophrenia. One group will receive standard antipsychotic medication plus 60mg Raloxifene, the second group receives standard antipsychotic medication plus Hormone Therapy(estradiol 2mg oral per day + dyhydroprogesterone 10mg oral per day) and the third group receives standard antipsychotic medication plus oral placebo. Hypothesis 1: That the women receiving adjunctive raloxifene or HT would have a quicker recovery from psychotic symptoms, as measured on the rating scales, compared with the women receiving adjunctive placebo.Hypothesis 2: That the Raloxifene group would have better cognitive improvement than the other two groups.

DETAILED DESCRIPTION:
Estrogen is hypothesised to be protective for women against early onset of severe symptoms of schizophrenia (Hafner,1991; Seeman, 1992). This "estrogen hypothesis" was derived from epidemiological, clinical and animal studies. Following the results of such studies, we conducted a study (Kulkarni et al 1996) in which a group of premenopausal women with schizophrenia were given 0.02mg oral estradiol as an adjunct to antipsychotic drug treatment for 8 weeks and compared their progress with a similar group who received antipsychotic drugs only. The group receiving estrogen made a significantly more rapid recovery from acute psychotic symptoms and also reported improvement in their general health status. Subsequently, we have conducted a 4 week double blind, placebo controlled study using 100 microgram estradiol skin patch. We found that the 12 pre-menopausal women who received the estradiol adjunct had a significantly lower total PANSS and BPRS score than 12 women who received placebo patches plus antipsychotic medication. (Kulkarni et al 2000).

The major potential risks in using estrogen as a longer-term adjunctive treatment in pre-menopausal women with schizophrenia appear to be the potential harmful effects of estrogen itself in its action on breast and uterine tissue. Our studies were brief for this reason, in that we used estrogen without progesterone over an 8 week or 4 week period.

With the recent advent of selective estrogen receptor modulators, in particular raloxifene hydrochloride, there is the potential to harness the positive estrogenic effect on CNS neurotransmitter systems without affecting breast or uterine tissue. While the CNS effects of raloxifene have not been fully studied, its actions are mediated through binding to estrogen receptors and can thereby regulate gene expression that is ligand, tissue or gene specific. By inference then, raloxifene would be expected to impact on dopamine and serotonin pathways in a similar fashion to conjugated estrogen. A study (Nickleisen et al 1999) on the effect of raloxifene on cognition in healthy, postmenopausal women found a slight increase in verbal memory performance after one month of high dose treatment, while no other differences were found after 12 months of treatment. There are no studies in women with cognitive impairment where a treatment effect would be more likely to be apparent. Similarly, there are no clinical studies to date investigating the effect of raloxifene on psychotic symptoms. To this end, we are putting forward an investigator initiated clinical trial proposal to investigate the effect of adjunctive raloxifene on psychotic symptoms in women with schizophrenia.

The aim of this project is to study the effect of raloxifene as an adjunct to antipsychotic medication in postmenopausal women with schizophrenia as a means of developing a novel, safe adjunctive treatment for women with schizophrenia to improve their quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Female aged over 45 years
* Current diagnosis of DSM-IV Schizophrenia, Schizoaffective or Schizophreniform Disorder
* Symptom rating greater than 60 on the PANSS at baseline/screening
* Patient able to give informed consent
* Patient post menopausal (confirmed by hormone assay and Greene Climacteric Scale plus Menstrual Cycle Questionnaire)

Exclusion Criteria:

* Clinically significant concomitant medical or neurological condition or history of venous thromboembolic event
* High suicide/aggression Risk in the opinion of the investigator.
* If patient's psychotic illness is directly related to illicit substance abuse or has a history of substance abuse or dependence in the past 6 months
* Smoking more than 20 cigarettes per day
* Use of any form of hormones or hormone therapy
* Illness causing immobilisation
* Undiagnosed postmenopausal vaginal bleeding
* Consumption of more than 30gm of alcohol (3 standard drinks)per day.

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2002-10; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
PANSS score at trial completion (12 weeks)

SECONDARY OUTCOMES:
MADRS score at trial completion (12 weeks)
Cognitive Test scores at trial completion (12 weeks)
Adverse Symptom Checklist score at trial completion (12 weeks)
Hormone level change over study period (12 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Jayashri Kulkarni, MBBS, MPM, FRANZCP, PHD, Principal Investigator — Bayside Health; Alfred Hospital
Locations (1):
- Alfred Psychiatry Research Centre, Alfred Hospital, Melbourne, Victoria, Australia